CLINICAL TRIAL: NCT06326281
Title: Comparison of External Oblique Intercostal Plane Block Oblique Subcostal Transversus Abdominis Plane Block and Local Anesthetic Infiltration Methods in Laparoscopic Cholecystectomies
Brief Title: Postoperative Pain Management in Laparoscopic Cholecystectomies
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Selahattin Buğra Kurtoğlu, Assistant doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACHBILKENT-ANEST-BK-01
Record Dates: First submitted 2024-03-17; First posted 2024-03-22 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Postoperative Pain; Regional Anesthesia
Keywords: regional anesthesia; laparoscopic cholecystectomy; external oblique intercostal plane block; postoperative pain; analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Control Groups; Tramadol

STUDY DESIGN:
Intervention Model Description: Evaluation of postoperative pain in 4 groups in laparoscopic cholecystectomy with control group
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients were not told which method would be used The person evaluating the patients did not know which method was applied to which patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- External oblique intercostal plane block group (Active Comparator): Before general anaesthesia, Ultrasound guided unilateral external oblique intercostal plane block group block will perform with 20 ml of 0.25% bupivacaine .Patient controlled analgesia with tramadol will apply to the all patients. Postoperative pain assessment and opioid consumption will record till the postoperative 24 th hours.
  Interventions: Procedure: unilateral external oblique intercostal plane block group
- Oblique subcostal transversus abdomınıs plane block group (Active Comparator): Under general anaesthesia, Ultrasound guided unilateral oblique subcostal transversus abdomınıs plane block will perform with 20 ml of 0.25% bupivacaine. Patient controlled analgesia with tramadol will apply to the all patients. Postoperative pain assessment and opioid consumption will record till the postoperative 24 th hours
  Interventions: Procedure: unilateral oblique subcostal transversus abdomınıs plane block group
- Local anesthetic infiltration group (Active Comparator): 4 trocars will be used by the surgical team during the operation, and these trocars will be placed 10 mm infraumbilical, 10 mm in the middle epigastrium, 5 cm below the xiphoid, 5 mm in the midclavicular line and in the right subcostal region, and 5 mm in the anterior axillary line. Before trocar placement, 0.25% bupivacaine will be applied to the skin, fascia, muscle and preperitoneal area in accordance with the infiltration rules. A total of 20 mL of 0.25% bupivacaine will be used, 6 mL for 10 mm trocar sites and 4 mL for 5 mm trocar sites. Patient controlled analgesia with tramadol will apply to the all patients. Postoperative pain assessment and opioid consumption will record till the postoperative 24 th hours
  Interventions: Procedure: Local anesthetic infiltration group
- Control Group (Sham Comparator): All patients were followed using a standardized postoperative analgesia protocol which includes tramadol patient controlled analgesia. Tramadol at a concentration of 5 mg/mL is included in our patient controlled analgesia protocol (total volume 100 mL.) Patient controlled analgesia protocols were set to no basal infusion and 10 mg bolus doses with a 20 min lock time 25 patient included and patients were observed for pain for 24 hours
  Interventions: Drug: Control group

INTERVENTIONS:
Procedure: unilateral external oblique intercostal plane block group — USG guided external oblique intercostal plane block will perform unilateral with Bupivacaine 25 patient included and patients were observed for pain for 24 hours
  Arms: External oblique intercostal plane block group
Procedure: unilateral oblique subcostal transversus abdomınıs plane block group — USG guided oblique subcostal transversus abdomınıs plane block block will perform unilateral with Bupivacaine. 25 patient included and patients were observed for pain for 24 hours
  Arms: Oblique subcostal transversus abdomınıs plane block group
Procedure: Local anesthetic infiltration group — Bupivacaine infiltration will be performed to trocar insertion sites. 25 patient included and patients were observed for pain for 24 hours
  Arms: Local anesthetic infiltration group
Drug: Control group — All patients were followed using a standardized postoperative analgesia protocol which includes tramadol patient controlled analgesia. Tramadol at a concentration of 5 mg/mL is included in our patient controlled analgesia protocol (total volume 100 mL.) patient controlled analgesias were set to no basal infusion and 10 mg bolus doses with a 20 min lock time 25 patient included and patients were observed for pain for 24 hours
  Other Names: intravenous patient controlled analgesia group with tramadol
  Arms: Control Group

SUMMARY:
This study is to demonstrate the effectiveness of external oblique intercostal plane block, a new block method, in the treatment of postoperative pain occurring after laparoscopic cholecystectomy operations, which are frequently and widely performed today.

It aims to add new applications to multimodal analgesia methods, which provide the greatest contribution to the early recovery process after surgery, and to contribute to the early recovery process by increasing patient satisfaction.

DETAILED DESCRIPTION:
Postoperative pain is an acute pain that begins with surgical trauma and gradually decreases with tissue healing, and its elimination is important for ideal patient care after surgery. Postoperative pain; It varies depending on the type of surgery, the patient, and the need and type of analgesic in the intraoperative period. Although there have been new developments in recent years to relieve postoperative pain, studies have shown that 25% of patients can receive adequate postoperative pain treatment.The increase in thromboembolic, cardiac and respiratory complications caused by untreatable postoperative pain is one of the most important problems in operated patients.

Laparoscopic cholecystectomy; It is one of the most frequently performed surgical procedures in adult patients, and different types of pain such as parietal, visceral and somatic (shoulder pain) can be observed due to tissue damage after laparoscopic cholecystectomy, postoperative pain, diaphragmatic irritation and residual pneumoperitoneum.Multimodal analgesia in laparoscopic cholecystectomies; It can be provided with combinations of regional anesthesia techniques, incision site local anesthetic applications, intravenous opioids, nonsteroidal anti-inflammatory drugs, paracetamol and preemptive analgesia methods.

Regional anesthesia techniques have become more popular recently for the purpose of postoperative pain control, and regional anesthesia techniques in laparoscopic cholecystectomy such as epidural block, paravertebral block, transversus abdominis plan (TAP) block and External Oblique Intercostal Plan (EOIP) block, whose effectiveness has been shown by new studies. Includes methods.

Oblique subcostal transversus abdominis plane (OSTAP) block is a regional anesthesia technique defined as a modified version of the TAP block used especially in upper abdominal surgeries such as Laparoscopic cholecystectomy.EOIP block is a new regional anesthesia technique that can provide analgesia in the postoperative period in upper abdominal abdominal surgery, which was demonstrated by anatomical studies in 2021.

EOIP block, the spread of regional anesthesia to the lateral and anterior cutaneous branches of T6/7 and T10/11, the origin of the intercostal nerves, constitutes the mechanism of this technique and shows that Laparoscopic cholecystectomies can be effective in postoperative analgesia management.

Regional anesthesia methods are frequently used in our clinic for patients undergoing upper abdominal surgery for analgesia. In this study, the investigators aimed to compare the EOIP block, OSTAP block and local anesthetic infiltration methods in laparoscopic cholecystectomy in terms of pain effectiveness in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65
* Patients undergoing elective laparoscopic cholecystectomy
* American Society of Anesthesiologists score 1-2 patients
* Body mass index ) <35kg/m2
* Patients whose consent was obtained before the procedure

Exclusion Criteria:

* Patients under the age of 18 and over the age of 65
* American Society of Anesthesiologists score III and above
* Surgeries with an operating time exceeding 120 minutes
* Emergency surgeries
* Those who have had abdominal surgery
* Pregnant or breastfeeding patients
* Those who have coagulopathy and use anticoagulant drugs
* Those who are allergic to local anesthetics
* Those with localized infection at the injection site
* Patients who do not have the ability to use patient controlled analgesia and evaluate Numerical rating scale
* Patients with peripheral nerve disease
* Patients with renal failure and congestive heart failure
* Patients undergoing elective laparoscopic cholecystectomy due to malignancy
* Surgeries where open surgery is performed during the operation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
Amount of postoperative opioid use | 24 hours
  Patient controlled analgesia (PCA) will provide with tramadol PCA. Total tramadol consumption will calculate and record till the postoperative 24th hours
Finding out which method is more effective according to the Numerical Rating Scale (0-10) | 24 hours
  To find out which method provides more effective analgesia according to the Numeric Rating Scale patients followed for 24 hours. A numerical rating scale (NRS) requires the patient to rate their pain on a defined scale.
  0 is no pain and 10 is the worst pain

SECONDARY OUTCOMES:
postoperative nause and vomiting | 24 hours
  The patient with nausea and vomiting will be recorded
  postoperative nausea and vomiting; will be evaluated as present or absent
postoperative shoulder pain | 24 hours
  The patient with shoulder pain will be recorded
  postoperative shoulder pain; will be evaluated as present or absent

CONTACTS AND LOCATIONS:
Overall Officials: Buğra Kurtoğlu, MD, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bılkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No